CLINICAL TRIAL: NCT03576755
Title: Pilot Randomized Controlled Trial of Spironolactone in Young Women With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Spironolactone Therapy In Young Women With NASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18-24453
Record Dates: First submitted 2018-04-18; First posted 2018-07-03 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Canrenoic Acid

STUDY DESIGN:
Intervention Model Description: The following treatment regimens will be used:
  * Experimental treatment - spironolactone, 100 mg once daily
  * Placebo or Comparator - one capsule, once daily
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, research staff, or patients. The following study procedures will be in place to ensure double-blind administration of study treatments Access to the randomization code will be strictly controlled. A color and size-matched placebo capsule that looks identical to the spironolactone capsule will be used.
  Packaging and labeling of test and control treatments will be identical to maintain the blind.
  The study blind will be broken on completion of the clinical study, after all study endpoints have been ascertained by blinded study coordinators and after the study database has been locked.
  During the study, the blind may be broken only in emergencies when knowledge of the patient's treatment group is necessary for further patient management. The UCSF investigational pharmacy would then be notified and responsible for unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- spironolactone (Experimental): spironolactone, 100 mg capsule administered orally once daily for 6 or 12 months
  Interventions: Drug: Spironolactone 100mg
- placebo (Placebo Comparator): matching placebo capsule administered orally once daily for 6 or 12 months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Spironolactone 100mg — Spironolactone capsules will be prepared from USP grade powder at a dose of 100 mg.
  Arms: spironolactone
Drug: Placebo oral capsule — Matching placebo capsules of the same color, mass, and appearance to the spironolactone capsules will be filled using microcrystalline cellulose powder.
  Arms: placebo

SUMMARY:
Nonalcoholic steatohepatitis (NASH), or fat-related liver inflammation and scarring is projected to be the leading cause of cirrhosis in the United States (U.S.) within the next few years. Women are at disproportionate risk for NASH, with approximately 15 million U.S. women affected. There is an urgent need to understand risk factors for NASH and its progression in women, and sex hormones may provide a missing link.

The investigator's preliminary data support a detrimental role of androgens, or "male sex hormones" on fatty liver in women but no studies have evaluated whether androgens are associated with liver inflammation and/or scarring from fatty liver (aka NASH). To better understand the mechanism by which androgens might promote NASH and/or metabolic co-factors that contribute to NASH, the investigators are conducting a pilot clinical trial to primarily assess the feasibility of using an androgen blocking medication, spironolactone, in women with NASH. Spironolactone was selected because it is has been commonly prescribed for decades with good safety profile and tolerability to treat symptoms of high androgens, like acne and hirsutism in young women. Though primarily a feasibility-focused study, the investigators also aim to explore the pathways by which blocking testosterone receptors might alter the biologic processes that promote NASH and its associated metabolic co-morbidities in women.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized, (2:1) parallel group pilot clinical trial of spironolactone in women with biopsy-proven NASH receiving 6 or 12 months of spironolactone or placebo. 30 women are targeted for enrollment. Each participant will be administered a single dose of spironolactone or placebo once daily for a total of 6 or 12 months. In person evaluations will take place at Month 1, 3, 6, 9, and 12. There will be a telephone follow up visit within 3 months of end of treatment (up to Month 9 or 15).

This is a pilot clinical trial that is largely feasibility focused. Study outcomes will include

* Change in liver stiffness on Magnetic Resonance Elastography (MRE)
* Change in hepatic steatosis by Magnetic Resonance Proton Density Fat Fraction (PDFF)
* Change in visceral adipose tissue (VAT) volume by Magnetic Resonance Imaging (MRI)
* Change in NASH histology as assessed by the continuous NAFLD activity score (NAS), which measures different components of NASH on liver biopsy.
* Biochemical endpoints: serum lipids & HOMA-IR
* Feasibility outcomes including Rates (and reasons) for the following: a) % women that decline/women contacted for study inclusion (i.e. need for a second liver biopsy, concern regarding randomization to placebo) b) % women enrolled/women screened (i.e. exclusion criteria too narrow), c) study dropout (i.e. medication side effects, too frequent study visits, and/or phlebotomy)

ELIGIBILITY:
Inclusion Criteria:

1. Women 18-45 years of age at Baseline Visit.
2. Documentation of NASH diagnosis confirmed on baseline liver biopsy (performed as clinical care) prior to study enrollment.
3. Written informed consent (and assent when applicable) obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
3. Uncontrolled diabetes (HbA1c 9.5% or higher within 60 days prior to enrollment)
4. Routine alcohol consumption >7 drinks per week during the preceding 3 months prior to baseline liver biopsy.
5. Other forms of chronic liver disease including hepatitis B virus infection (hepatitis B surface antigen positive), chronic hepatitis C virus (HCV) infection (HCV Ab and HCV ribonucleic acid positive), autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, and autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, iron overload, and alpha-1-antitrypsin deficiency, based on medical history and/or centralized review of liver histology
6. Any prior or upcoming weight reduction surgery (e.g., Roux-en-Y or gastric bypass)
7. HIV infection
8. Receipt of drugs associated with NAFLD (i.e. amiodarone, methotrexate, systemic glucocorticoids, tamoxifen, anabolic steroids, valproic acid) for more than 4 weeks prior to baseline or between baseline and follow-up biopsies
9. Perimenopausal status (defined as within 3 years of self-reported menopause) due to unstable hormonal levels during that time
10. Renal impairment defined as glomerular filtration rate <45 ml/min/1.73m or potassium levels > 5.0 mmol/L due to the diuretic effect of spironolactone
11. Participation in another clinical trial of an investigational drug or device
12. History of medication non adherence as noted upon chart review or patient report of difficulty with medication adherence
13. Androgen receptor antagonist use (i.e. flutamine, spironolactone or flutamide) for more than 3 months within one year prior to baseline biopsy
14. Eplerenone use as this is a diuretic that also blocks the aldosterone receptor and could compound side effects
15. Cirrhosis on baseline biopsy as this condition leads to altered sex hormone metabolism
16. Unstable dosing (i.e. dose increase, intermittent use, or initiation) of Vitamin E anytime during the 3 months prior to baseline biopsy
17. Significant weight loss (at least 10% decrease in body weight) over preceding 3 months prior to baseline biopsy
18. Contraindication to MRI scanning (e.g. presence of permanent pacemakers, implanted cardiac devices, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika A Sarkar, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlton MR, Burns JM, Pedersen RA, Watt KD, Heimbach JK, Dierkhising RA. Frequency and outcomes of liver transplantation for nonalcoholic steatohepatitis in the United States. Gastroenterology. 2011 Oct;141(4):1249-53. doi: 10.1053/j.gastro.2011.06.061. Epub 2011 Jul 2. PMID 21726509
- [Background] Wong RJ, Cheung R, Ahmed A. Nonalcoholic steatohepatitis is the most rapidly growing indication for liver transplantation in patients with hepatocellular carcinoma in the U.S. Hepatology. 2014 Jun;59(6):2188-95. doi: 10.1002/hep.26986. Epub 2014 Apr 25. PMID 24375711
- [Background] Sarkar M, Wellons M, Cedars MI, VanWagner L, Gunderson EP, Ajmera V, Torchen L, Siscovick D, Carr JJ, Terry JG, Rinella M, Lewis CE, Terrault N. Testosterone Levels in Pre-Menopausal Women are Associated With Nonalcoholic Fatty Liver Disease in Midlife. Am J Gastroenterol. 2017 May;112(5):755-762. doi: 10.1038/ajg.2017.44. Epub 2017 Mar 14. PMID 28291240
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Bambha K, Belt P, Abraham M, Wilson LA, Pabst M, Ferrell L, Unalp-Arida A, Bass N; Nonalcoholic Steatohepatitis Clinical Research Network Research Group. Ethnicity and nonalcoholic fatty liver disease. Hepatology. 2012 Mar;55(3):769-80. doi: 10.1002/hep.24726. PMID 21987488
- [Background] Neuschwander-Tetri BA, Clark JM, Bass NM, Van Natta ML, Unalp-Arida A, Tonascia J, Zein CO, Brunt EM, Kleiner DE, McCullough AJ, Sanyal AJ, Diehl AM, Lavine JE, Chalasani N, Kowdley KV; NASH Clinical Research Network. Clinical, laboratory and histological associations in adults with nonalcoholic fatty liver disease. Hepatology. 2010 Sep;52(3):913-24. doi: 10.1002/hep.23784. PMID 20648476
- [Background] Kelley CE, Brown AJ, Diehl AM, Setji TL. Review of nonalcoholic fatty liver disease in women with polycystic ovary syndrome. World J Gastroenterol. 2014 Oct 21;20(39):14172-84. doi: 10.3748/wjg.v20.i39.14172. PMID 25339805
- [Background] Vassilatou E. Nonalcoholic fatty liver disease and polycystic ovary syndrome. World J Gastroenterol. 2014 Jul 14;20(26):8351-63. doi: 10.3748/wjg.v20.i26.8351. PMID 25024594
- [Background] Macut D, Tziomalos K, Bozic-Antic I, Bjekic-Macut J, Katsikis I, Papadakis E, Andric Z, Panidis D. Non-alcoholic fatty liver disease is associated with insulin resistance and lipid accumulation product in women with polycystic ovary syndrome. Hum Reprod. 2016 Jun;31(6):1347-53. doi: 10.1093/humrep/dew076. Epub 2016 Apr 12. PMID 27076501
- [Background] Lovejoy JC, Bray GA, Bourgeois MO, Macchiavelli R, Rood JC, Greeson C, Partington C. Exogenous androgens influence body composition and regional body fat distribution in obese postmenopausal women--a clinical research center study. J Clin Endocrinol Metab. 1996 Jun;81(6):2198-203. doi: 10.1210/jcem.81.6.8964851.
- [Background] Corbould A. Effects of androgens on insulin action in women: is androgen excess a component of female metabolic syndrome? Diabetes Metab Res Rev. 2008 Oct;24(7):520-32. doi: 10.1002/dmrr.872. PMID 18615851
- [Background] Croston GE, Milan LB, Marschke KB, Reichman M, Briggs MR. Androgen receptor-mediated antagonism of estrogen-dependent low density lipoprotein receptor transcription in cultured hepatocytes. Endocrinology. 1997 Sep;138(9):3779-86. doi: 10.1210/endo.138.9.5404. PMID 9275065
- [Background] Wada T, Kenmochi H, Miyashita Y, Sasaki M, Ojima M, Sasahara M, Koya D, Tsuneki H, Sasaoka T. Spironolactone improves glucose and lipid metabolism by ameliorating hepatic steatosis and inflammation and suppressing enhanced gluconeogenesis induced by high-fat and high-fructose diet. Endocrinology. 2010 May;151(5):2040-9. doi: 10.1210/en.2009-0869. Epub 2010 Mar 8. PMID 20211973

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients withdrew consent prior to randomization. All other participants were immediately randomized once baseline was completed.
Groups:
- Spironolactone 6: spironolactone, 100 mg capsule administered orally once daily for 6 months
  Spironolactone 100mg: Spironolactone capsules will be prepared from USP grade powder at a dose of 100 mg.
- Placebo 6: matching placebo capsule administered orally once daily for 6 months
  Placebo oral capsule: Matching placebo capsules of the same color, mass, and appearance to the spironolactone capsules will be filled using microcrystalline cellulose powder.
- Spironolactone 12: spironolactone, 100 mg capsule administered orally once daily for 12 months
  Spironolactone 100mg: Spironolactone capsules will be prepared from USP grade powder at a dose of 100 mg.
- Placebo 12: matching placebo capsule administered orally once daily for 12 months
  Placebo oral capsule: Matching placebo capsules of the same color, mass, and appearance to the spironolactone capsules will be filled using microcrystalline cellulose powder.
Period: Overall Study
Arm/Group | Spironolactone 6 | Placebo 6 | Spironolactone 12 | Placebo 12
Started | 3 | 4 | 8 | 2
Completed | 2 | 4 | 8 | 2
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 33 [18 to 44] | 30 [21 to 45] | 32 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 6 | 17
Diagnosed with PCOS [Count of Participants; unit: Participants] | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Stiffness on Magnetic Resonance Elastography (MRE)
Description: The investigators will assess for change in the MRE quantified liver stiffness in kilopascals (kPA)
Time Frame: 6 or 12 Months
Population: Median (IQR) change in kPA will be reported from baseline to 6 months and separately baseline to 12 months by treatment group.
Measure: Median (Inter-Quartile Range); unit: Change in kPA
Groups:
- Spironolactone 6: spironolactone, 100 mg capsule administered orally once daily for 6
  Spironolactone 100mg: Spironolactone capsules will be prepared from USP grade powder at a dose of 100 mg.
- Placebo 6: matching placebo capsule administered orally once daily for 6
  Placebo oral capsule: Matching placebo capsules of the same color, mass, and appearance to the spironolactone capsules will be filled using microcrystalline cellulose powder.
- Sprionolactone 12: spironolactone, 100 mg capsule administered orally once daily for 12
  Spironolactone 100mg: Spironolactone capsules will be prepared from USP grade powder at a dose of 100 mg.
- Placebo 12: matching placebo capsule administered orally once daily for 12
  Placebo oral capsule: Matching placebo capsules of the same color, mass, and appearance to the spironolactone capsules will be filled using microcrystalline cellulose powder.
Arm/Group | Spironolactone 6 | Placebo 6 | Sprionolactone 12 | Placebo 12
Number analyzed (Participants) | 10 | 6 | 8 | 3
Change in kPA | 0.025 [-0.330 to 0.350] | -0.265 [-0.340 to 0.090] | 0.105 [-0.035 to 0.770] | 0.135 [-0.220 to 0.490]

2. Secondary Outcome: Change in Hepatic Steatosis by Magnetic Resonance Proton Density Fat Fraction (PDFF)
Description: The investigators will assess for % change in fat fraction by MRI-PDFF
Time Frame: 6 or 12 months
Population: Standard error change in % will be reported from baseline to 6 months and separately baseline to 12 months by treatment group.
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Spironolactone 6 | Placebo 6 | Sprionolactone 12 | Placebo 12
Number analyzed (Participants) | 10 | 6 | 8 | 3
% change | -4.95 [-6.60 to 3.10] | -3.05 [-6.60 to 11.10] | -5.20 [-6.35 to -2.95] | -3.20 [-8.30 to 0.20]

3. Secondary Outcome: Change in Visceral Adipose Tissue (VAT) Volume by Magnetic Resonance Imaging (MRI)
Description: The investigators will assess for change in the MRI quantified VAT volume cm^2
Time Frame: 6 or 12 months
Population: Median (IQR) change in cm^2 will be reported from baseline to 6 months and separately baseline to 12 months by treatment group.
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Spironolactone 6 | Placebo 6 | Sprionolactone 12 | Placebo 12
Number analyzed (Participants) | 10 | 6 | 8 | 3
cm^2 | 3.3 [-4.4 to 9.6] | 11.9 [-5.2 to 12.9] | 6.8 [-7.4 to 16.8] | 18.3 [10.0 to 32.6]

4. Secondary Outcome: Change HOMA-IR (Homeostatic Model Assessment (HOMA) for Insulin Resistance (IR)).
Description: The investigators will assess change in continuous measures of HOMA-IR as insulin resistance is known to contribute to NASH progression. HOMA-IR was calculated as: Fasting serum insulin (mU/L) x Fasting plasma glucose (mmol/L) / 22.5. Higher scores indicate greater insulin resistance and a worse outcome. There is no theoretical minimum and/or maximum value for HOMA-IR.
Time Frame: 6 or 12 Months
Population: Median (IQR) change will be reported (mU/L*mmol/L) from baseline to 6 months and separately from baseline to 12 months by treatment group.
Measure: Median (Inter-Quartile Range); unit: mU/L*mmol/L
Arm/Group | Spironolactone 6 | Placebo 6 | Sprionolactone 12 | Placebo 12
Number analyzed (Participants) | 10 | 6 | 8 | 3
mU/L*mmol/L | 5.29 [3.46 to 14.30] | 4.49 [3.63 to 7.80] | 5.99 [3.43 to 7.30] | 11.90 [4.80 to 24.62]

5. Secondary Outcome: Change in the Non-Alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS 0-8).
Description: The investigators will assess for change in this histologic scoring system of NASH as a continuous measure among women willing to undergo end of treatment biopsy (not required). The NAS scoring is used to assess the severity and activity of NAFLD taking into account three components: steatosis (fat accumulation) scored from 0 to 3, Lobular inflammation scored from 0 to 3, and hepatocyte ballooning scored from 0 to 2. The total NAS score ranges from 0 to 8. Higher scores indicate greater disease activity. Interpretation of NAS scores: 0-2 no significant NAFLD, 3-4, borderline NASH, and 5-8, definite NASH. As this was an optional component of the study, none of the participants who completed 6 months chose to undergo the biopsy which is why we only have 12 month measurements.
Time Frame: 6 or 12 Months
Population: Median (IQR) change will be reported from baseline to 12 months by treatment group.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Sprionolactone 12 | Placebo 12
Number analyzed (Participants) | 3 | 2
scores on a scale | 2 [0 to 2] | 2.5 [2 to 3]

ADVERSE EVENTS:
Time Frame: Through study completion on average 1 year.
Arm/Group | Spironolactone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 6/11 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=11) | Placebo (N=6)
Polydipsia (General disorders) | 1 (1) | 1 (1) — Feeling of dry mouth
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — pt reported cramping 3 inches below right breast occurring for less than 10 seconds. In the middle of the night
Dark urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Right ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck stiffness/pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cough and sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Stomach cramping/abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Lightheadeness (General disorders) | 0 (0) | 1 (1)
Fatigue/ increased fatigue (General disorders) | 1 (1) | 3 (3)
Fever (Immune system disorders) | 0 (0) | 2 (3)
Worsened bilateral otalgia/otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)
nasal congestion, sneezing, and rhinorrhea (Immune system disorders) | 1 (1) | 1 (1)
Increased anxiety/depression (Psychiatric disorders) | 0 (0) | 1 (1)
trigger finger of right hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Increased urination (Renal and urinary disorders) | 2 (2) | 1 (1)
eye twitching (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Herpes (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
bilateral hand itchiness (General disorders) | 1 (1) | 0 (0)
shoulder and abdominal pain after biopsy (Surgical and medical procedures) | 1 (1) | 0 (0)
amenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
COVID-19 infection (Infections and infestations) | 0 (0) | 1 (1)
Increased hair loss (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
left pinched nerve and neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03576755/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT03576755/ICF_001.pdf